CLINICAL TRIAL: NCT07175428
Title: A Phase 2, Randomized, Multicenter, Open-label, Blinded-endpoint Study to Evaluate the Safety of REGN7508 and REGN9933, Monoclonal Antibodies Against FXI, Versus Apixaban in Participants With Atrial Fibrillation (ROXI-ATLAS)
Brief Title: Safety in Adult Participants With Atrial Fibrillation Who Are Treated With Anticoagulation
Acronym: ROXI-ATLAS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R7508-CVA-2393
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Atrial Fibrillation (AF)
Keywords: Bleeding; Stroke; Systemic embolism; Blood clots
MeSH Terms: conditions — Atrial Fibrillation; Hemorrhage; Stroke; Thrombosis | interventions — apixaban

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- REGN7508 (Experimental)
  Interventions: Drug: REGN7508
- REGN9933 (Experimental)
  Interventions: Drug: REGN9933
- Apixaban (Active Comparator)
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: REGN7508 — Administered per the protocol
  Arms: REGN7508
Drug: REGN9933 — Administered per the protocol
  Arms: REGN9933
Drug: Apixaban — Administered per the protocol
  Other Names: Eliquis
  Arms: Apixaban

SUMMARY:
This study is researching experimental drugs called REGN7508 and REGN9933. The study is focused on participants who have atrial fibrillation, which means that the heart beats too fast and unevenly. REGN7508 and REGN9933 are designed to help stop blood clots forming in patients with atrial fibrillation.

The aim of the study is to see how well REGN7508 and REGN9933 work in patients that get medicine for their atrial fibrillation. The bleeding effects of REGN7508 and REGN9933 will be compared to another medicine (apixaban), which is available on the market to treat and prevent formation of blood clots.

The study is looking at several other research questions, including:

* What side effects may happen from taking REGN7508 or REGN9933
* How well do the study drugs reduce the risk of having a stroke
* How much of REGN7508 or REGN9933 is in the blood at different times
* Whether the body makes antibodies against REGN7508 or REGN9933 (which could make the drugs less effective or could lead to side effects)

ELIGIBILITY:
Key Inclusion Criteria:

1. Has AF or flutter (paroxysmal or persistent), not felt to be secondary to a reversible cause, and an indication for indefinite anticoagulation treatment as described in the protocol
2. Meets one of the following:

   1. CHA2DS2-VA [C: Congestive heart failure; H: Hypertension; A2: Age ≥75 years (double points); D: Diabetes mellitus; S2: Stroke or TIA or Thromboembolism (double points); V: Vascular disease; A: Age 65-74 years] score ≥2 and Oral Anticoagulant (OAC) naïve or
   2. CHA2DS2-VA score ≥3 or
   3. CHA2DS2-VA score of 2 and at least 1 enrichment criteria as described in the protocol
3. Must have a Prothrombin Time/International Normalization Ratio (PT/INR) <2.5 at the time of randomization if taking warfarin or another Vitamin K Antagonist (VKA)

Key Exclusion Criteria:

1. Has a mechanical heart valve prosthesis (Note: transcatheter aortic valve replacement is not an exclusion)
2. Has known moderate-to-severe mitral stenosis
3. Has had successful ablation therapy or Left Atrial Appendage (LAA) occlusion/exclusion, or planned ablation or LAA occlusion/exclusion as described in the protocol
4. Had an ischemic stroke within 2 days prior to randomization
5. Has Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) estimated Glomerular Filtration Rate (eGFR) <15 mL/min/1.73m^2 within 14 days prior to randomization or on dialysis or expected to be started as described in the protocol
6. Has a history of central nervous system bleeding within 30 days prior to randomization

Note: Other protocol-defined Inclusion/ Exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2027-02-09 (Estimated); Study Completion 2027-04-21 (Estimated)

PRIMARY OUTCOMES:
Incidence of any bleeding | 12 weeks
  Defined as the composite of International Society on Thrombosis and Haemostasis (ISTH) major bleeding, ISTH Clinically Relevant Non-Major (CRNM) bleeding, or minor bleeding

SECONDARY OUTCOMES:
Incidence of the composite of ISTH major bleeding or ISTH CRNM bleeding | 12 weeks
Incidence of ISTH major bleeding | 12 weeks
Incidence of ISTH CRNM bleeding | 12 weeks
Incidence of minor bleeding | 12 weeks
Number of ISTH major bleeding events | 12 weeks
Number of ISTH CRNM bleeding events | 12 weeks
Number of minor bleeding events | 12 weeks
Incidence of Treatment-Emergent Adverse Events (TEAEs) | Approximately 25 weeks
Severity of TEAEs | Approximately 25 weeks
Incidence of the composite of stroke or systemic embolism | Approximately 12 weeks
Incidence of Antidrug Antibodies (ADA) to REGN7508 | 12 weeks
Magnitude of ADA to REGN7508 | 12 weeks
Incidence of ADA to REGN9933 | 12 weeks
Magnitude of ADA to REGN9933 | 12 weeks
Concentrations of REGN7508 | Approximately 25 weeks
Concentrations of REGN9933 | Approximately 25 weeks
Change from baseline in activated Partial Thromboplastin Time (aPTT) | Approximately 25 weeks
Change from baseline in Prothrombin Time (PT) | Approximately 25 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (25):
- United States (25):
  - SEC Clinical Research, Dothan, Alabama
  - Eastern Shore Research Institute, Fairhope, Alabama
  - Mission Cardiovascular Research Institute, Fremont, California
  - National Institute of California Heart and Vein Specialists, Huntington Beach, California
  - Profound Research LLC at Southern California Heart Specialists, Pasadena, California
  - Empire Clinical Research, Pomona, California
  - Cardiology Associates Medical Group, Ventura, California
  - Interventional Cardiology Medical Group, West Hills, California
  - Nouvelle Clinical Research LLC, Cutler Bay, Florida
  - Inpatient Research Clinic LLC, Miami Lakes, Florida
  - Cardiovascular Center of Sarasota Foundation for Research and Education, Sarasota, Florida
  - Clinical Site Partners, LLC DBA Flourish Research, Winter Park, Florida
  - NSC Research, Inc, Johns Creek, Georgia
  - Blue Coast Research Center, LLC, Indianapolis, Indiana
  - Franciscan Physician Network, Indiana Heart Physicians, Indianapolis, Indiana
  - Reid Physician Associates, Richmond, Indiana
  - Monroe Research, LLC, West Monroe, Louisiana
  - Anderson Medical Research, Ft. Washington, Maryland
  - Profound Research LLC, Farmington Hills, Michigan
  - AA Medical Research Center (MRC), Flint, Michigan
  - K&R Research LLC, Marion, Ohio
  - East Coast Institute for Research, Jefferson City, Jefferson City, Tennessee
  - PharmaTex Research, Amarillo, Texas
  - Tyler Cardiovascular Consultants, Tyler, Texas
  - Alpine Research TC, Clinton, Utah

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/